CLINICAL TRIAL: NCT00964535
Title: Bioequivalence Study Comparing Two Budesonide/Formoterol Fumarate Dihydrate Device-metered Dry Powder Inhalers, Budesonide/Formoterol Easyhaler 200/6 µg/Inhalation and Symbicort Turbohaler 200 µg/6 µg/Inhalation
Brief Title: Bioequivalence Study of Budesonide/Formoterol Easyhaler and Symbicort Turbohaler in Asthmatics
Acronym: KINECO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Ulla Sairanen, Orion Corporation, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3103002
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Budesonide/formoterol Easyhaler (Experimental)
  Interventions: Drug: budesonide and formoterol 200/6 microg
- Charcoal and Budesonide/formoterol EH (Experimental)
  Interventions: Drug: budesonide and formoterol 200/6 microg
- Symbicort Turbohaler (Active Comparator)
  Interventions: Drug: budesonide and formoterol 200/6 microg
- Charcoal and Symbicort Turbohaler (Active Comparator)
  Interventions: Drug: budesonide and formoterol 200/6 microg

INTERVENTIONS:
Drug: budesonide and formoterol 200/6 microg — 2 inhalations as a single dose
  Other Names: Budesonide/formoterol Easyhaler 200/6 microg/inhalation
  Arms: Budesonide/formoterol Easyhaler
Drug: budesonide and formoterol 200/6 microg — 2 inhalations as a single dose
  Other Names: Symbicort Turbohaler 200/6 microg/inhalation
  Arms: Symbicort Turbohaler
Drug: budesonide and formoterol 200/6 microg — 2 inhalations as a single dose with the concurrent charcoal blockage
  Other Names: Budesonide/formoterol Easyhaler 200/6 microg/inhalation
  Arms: Charcoal and Budesonide/formoterol EH
Drug: budesonide and formoterol 200/6 microg — 2 inhalations as a single dose with the concurrent charcoal blockage
  Other Names: Symbicort Turbohaler 200/6 microg/inhalation
  Arms: Charcoal and Symbicort Turbohaler

SUMMARY:
The purpose of this study is to compare the test product Budesonide/formoterol Easyhaler with the marketed product Symbicort Turbohaler in terms of the drug absorbed into the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-60 years with documented diagnosis of asthma
* Prebronchodilator forced expiratory volume in one second (FEV1) at least 80% of the predicted value
* The asthma should be stable on the same regular treatment for at least 4 weeks before screening.

Exclusion Criteria:

* Use of oral, parenteral or rectal corticosteroids within 4 weeks preceding the screening
* Respiratory infection within 4 weeks preceding the screening
* Any condition requiring regular concomitant treatment or likely to need concomitant treatment during the study with medicinal products which have pharmacokinetic interactions with budesonide
* Any disorder or clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters Cmax and AUCt of plasma budesonide and formoterol concentrations | within 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Sairanen, MSc, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom